CLINICAL TRIAL: NCT06133647
Title: Demographics, Characteristics and Outcomes of Male Breast Cancer Patients at Methodist Health System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 015.MTP.2023.A
Record Dates: First submitted 2023-07-06; First posted 2023-11-15 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Ductal Carcinoma in Situ; Invasive Lobular Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: managing Male Breast Cancer Patients at Methodist Health System — To determine the number of MBC cases as well as the demographics, characteristics, and outcomes of MBC patients at Methodist Health System (MHS).
  Other Names: Larger studies in MBC are needed to provide more clinical data to help guide treatment.

SUMMARY:
To determine the number of MBC cases as well as the demographics, characteristics, and outcomes of MBC patients at Methodist Health System (MHS).

DETAILED DESCRIPTION:
Male breast cancer (MBC) is a rare disease without sufficient clinical data supporting the management and treatment. The treatment of MBC arises from data extrapolated from female breast cancer (FBC). MBC has higher mortality than FBC. Previous studies have suggested differences between MBC and FBC; however, treatments remain the same for both. Larger studies in MBC are needed to provide more clinical data to help guide treatment.

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 18 years of age Patients diagnosed with ductal carcinoma in situ or invasive lobular carcinoma of the breast

Exclusion Criteria:

* 18 years of age

  * Prisoners
  * Pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * ≥ 18 years of age
  * Patients diagnosed with ductal carcinoma in situ or invasive lobular carcinoma of the breast
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
Diagnosis Rates of patients with MBC and FBC | 13 years
  complications of treatment
Recurrence rates of Patients with MBC and FBC | 13 years
  Recurrence rates of Patients with MBC and FBC
Duration of remission in Patients with MBC and FBC | 13 years
  Duration of remission in Patients with MBC and FBC
The Overall Survival of patients with MBC and FBC after receiving treatment | 13 years
  The Overall Survival of patients with MBC and FBC after receiving treatment
Determine the complications of Treatment in patients with MBC and FBC | 13 years
  Determine the complications of Treatment in patients with MBC and FBC

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute at Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes